CLINICAL TRIAL: NCT00462787
Title: A Phase I Dose Escalation Trial of Clofarabine in Addition to Topotecan, Vinorelbine, Thiotepa, and Dexamethasone in Pediatric Patients With Relapsed or Refractory Acute Leukemia
Brief Title: Combination Chemotherapy in Treating Young Patients With Relapsed or Refractory Acute Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-012; MSKCC-07012
Record Dates: First submitted 2007-04-18; First posted 2007-04-19 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-11

CONDITIONS: Leukemia
Keywords: acute undifferentiated leukemia; recurrent childhood acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Biphenotypic, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute | interventions — Filgrastim; Clofarabine; Dexamethasone; Thiotepa; Topotecan; Vinorelbine

ARMS (1):
- Clofarabine (Experimental): This is a single arm phase I clinical trial to assess safety (morbidity and mortality) of a novel leukemia re-induction regimen. The first component of this trial is a phase I dose escalation study to determine the maximum tolerated dose (MTD) of the novel agent Clofarabine, when used in combination with topotecan, vinorelbine, thiotepa and dexamethasone. A total of three dose levels will be explored in this study.
  Interventions: Biological: filgrastim; Drug: clofarabine; Drug: dexamethasone; Drug: thiotepa; Drug: topotecan hydrochloride; Drug: vinorelbine tartrate

INTERVENTIONS:
Biological: filgrastim
Drug: clofarabine
Drug: dexamethasone
Drug: thiotepa
Drug: topotecan hydrochloride
Drug: vinorelbine tartrate

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as clofarabine, topotecan, vinorelbine, thiotepa, and dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells.

PURPOSE: This phase I trial is studying the side effects and best dose of clofarabine when given together with topotecan, vinorelbine, thiotepa, and dexamethasone in treating young patients with relapsed or refractory acute leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of clofarabine when administered in combination with topotecan hydrochloride, vinorelbine ditartrate, thiotepa, and dexamethasone in young patients with relapsed or refractory acute leukemia.
* Evaluate the antileukemic potential of this regimen in these patients.
* Evaluate the incidence and severity of treatment-related morbidity and mortality in patients treated with this regimen.
* Develop a new reinduction treatment regimen that will result in a patient clinical response with as little residual disease as possible to permit a bone marrow transplantation while in subsequent remission; maintain the response long enough to identify an appropriate stem cell donor; and permit the patient to undergo a stem cell transplantation free of infections and without vital organ dysfunction.

OUTLINE: This is a nonrandomized, prospective, dose-escalation study of clofarabine.

Patients receive topotecan hydrochloride IV continuously over 120 hours on days 0-4; vinorelbine ditartrate over 6-10 minutes on days 0, 7, and 14; thiotepa IV over 4 hours on day 2; clofarabine IV over 2 hours on days 3-7; and oral or IV dexamethasone 3 times daily on days 3 and 7-13 and then on day 3 only thereafter. Patients also receive filgrastim (G-CSF) subcutaneously once daily beginning on day 8 and continuing until blood counts recover. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of clofarabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 2 of 6 patients experience dose-limiting toxicity OR the dose preceding that at which 2 of 3 patients experience dose-limiting toxicity. At least 6 patients are treated at the MTD.

After completion of study treatment, patients are followed once a week for 4 weeks, twice a month for 6 months, and then once a month for 2 years.

PROJECTED ACCRUAL: A total of 23 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Must have 1 of the following diagnoses:

  * Acute lymphoblastic leukemia (ALL) meeting 1 of the following criteria:

    * Refractory to initial induction with two or more standard regimens
    * Relapsed < 24 months after first complete response on a high-risk protocol OR refractory to one standard reinduction regimen
    * Second or greater relapse
  * Acute myeloid leukemia, acute biphenotypic leukemia, or acute undifferentiated leukemia meeting 1 of the following criteria:

    * Refractory to initial induction
    * First or greater relapse
* Must have > 20% bone marrow blasts, or evidence of recurrent disease at an extramedullary site
* No symptomatic CNS disease

  * Patients with asymptomatic CNS disease are eligible with the approval of the principal investigator

PATIENT CHARACTERISTICS:

* Karnofsky performance status (PS) 70-100% OR Lansky PS 70-100%
* AST and ALT < 4 times upper limit of normal
* Bilirubin < 2.0 mg/dL (unless liver involvement)
* Creatinine within normal range for age OR creatinine clearance > 60 mL/min/1.73 m^2
* Adequate cardiac function (either asymptomatic with no prior risk factors, or if symptomatic, left ventricular ejection fraction > 50% at rest)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active uncontrolled viral, bacterial, or fungal infection

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior clofarabine
* More than 2 weeks since prior systemic chemotherapy

  * At least 7 days since prior chemotherapy for patients with rapidly progressive disease and recovered

Max Age: 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2007-04; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of clofarabine | 2 years
Overall survival | 2 years
Progression-free survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter G. Steinherz, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Neerav Shukla, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States